CLINICAL TRIAL: NCT02647450
Title: An Exploratory Assessment of the Cost Impact of Managing GI Consequences of Cancer Treatment Outside of a Specialist Clinic
Brief Title: GI Consequences Economic Evaluation
Acronym: GICEE
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR 4447
Record Dates: First submitted 2016-01-05; First posted 2016-01-06 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GIANT Clinic Group: Patients are required to have been refereed to the GI and Nutrition team Clinic at the Royal Marsden Hospital. In the clinic they will be assessed for their symptoms using the Gastrointestinal Symptom Rating Scale (GSRS).
  Interventions: Other: GIANT Completed patient

INTERVENTIONS:
Other: GIANT Completed patient — Patients identified in the GIANT clinic and who fulfill the inclusion criteria will be sent a 9 page questionnaire. Upon receipt the questionnaire will be sent to the patient's GP for validation.

SUMMARY:
An estimated 90,000 patients are suffering from long term gastrointestinal problems after cancer treatments, and whilst the National Cancer Survivorship Initiative have been working to develop specific pathways of care, these pathways lack in both specialised tariff funding and awareness. This study aims to assess the economic and personal impact on patients suffering from stomach and/or bowel problems after cancer treatment prior to referral to the Gastrointestinal and Nutrition Team (GIANT) at the Royal Marsden Hospital. All patients referred to the GIANT service (including private patients but excluding re referrals) will be offered participation in the study.

The study will consist of a 9 page patient retrospective questionnaire, asking questions about investigations and medications prescribed over the past year, as well as costs and methods of trying to treat their symptoms themselves, and the personal cost to themselves of their symptoms through loss of work and emotional impact. As this questionnaire asks patients questions about the past year, and thus can be difficult to answer accurately, patient answers will be validated for reliability by sending a 1 page questionnaire to their GP asking the same questions about clinic visits concerning stomach/bowel problems, investigations and medications prescribed in the past year. Once this data is collected from the participants, and the study has finished, the average cost of clinical interventions, economic impact, and personal impact, will be calculated.

The results from this study will be useful in helping to show the economic burden of GI symptoms, and will provide evidence as to the economic benefit of specialised clinics for the consequences of cancer treatment; highlighting the need for a nationally recognised algorithm for management.

DETAILED DESCRIPTION:
The number of people who survive cancer has tripled in the past 30 years; however, chronic physical consequences of treatment for cancer adversely affect the quality of life of 20-25% of survivors. The largest group of patients reporting debilitating chronic side effects are those treated with radiotherapy alone or in combination with other treatments for pelvic cancer. Gastrointestinal symptoms are the most common chronic physical side effects reported, and have the greatest effect on daily activity. Overall, 50% of patients report that that their gastrointestinal symptoms affect their quality of life, and 20-40% state that this effect is moderate or severe. Such problems include chronic faecal incontinence (up to 60% of patients) after radiotherapy for prostate or rectal cancer (53, 54), and chronic loose stool (47%), defaecatory urgency (29%), or chronic abdominal pain (17%) after radiotherapy for gynecological cancer.

In 2010, the UK National Cancer Survivorship Initiative Vision challenged professionals to develop new models of care for patients because "the needs of cancer survivors are not being met, that being 'cured' of cancer does not necessarily equate with being well and that chronic consequences of treatment can have a devastating impact on daily life". The National Cancer Survivorship Initiative accepts that currently there is limited access to specialist services, despite an estimated 90,000 people in the UK experiencing long-term gastrointestinal problems as a consequence of cancer treatment. Furthermore, recent surveys of clinical oncologists and gastroenterologists concur with this sentiment, highlighting a lack of available expertise; with two UK audits of gastroenterology consultants and oncologists demonstrating no improvement in provision of specialist services between 2003 to 2010. Whilst NHS Improvement has developed stratified pathways of care, the Roadmap for Recovery report created recently by the Anthony Nolan Bone Marrow Transplant charity underlined the ongoing issue of lack of specialised commissioning of services for complex consequences of cancer treatment. It is estimated that £40 million (DoH) is wasted annually in futile and dangerous treatments for Pelvic Radiation Disease alone; academic estimates suggest this is closer to £80 million . Furthermore the incapacitating affects of GI symptoms leads to both loss of productivity and huge social costs. Currently there is no NHS tariff payable for GI consequences of cancer treatment; however the mean cost per completed episode of care by the GIANT (Gastrointestinal and Nutrition Team) service was calculated, amounting to an average cost of £1563 per patient. This can be compared to a tariff of £14,800 per woman treated with chemo-radiation for cervical cancer, and a cost in excess of £45,000 for a person with rectal cancer treated with long course chemo-radiation followed by surgery and adjuvant chemotherapy. With specialist clinics lacking, it can be assumed that the majority of people living with GI consequences of cancer treatment are being treated by their GPs; however, the Quality and Outcomes Framework by which GP Surgeries are measured and awarded financial incentives includes no domain or measure for gastrointestinal problems; and there have been no studies into the cost of managing patients with GI problems as a consequence of cancer treatment outside of the GIANT service. This exploratory study is a step in this direction.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* Past history of malignant disease.
* They are able to give informed consent to participate.
* Patients with longer term consequences of cancer treatment, defined as patients with symptoms referred 3 months or more after the end of their cancer treatment.

Exclusion Criteria:

* They have been re-referred to the GIANT clinic, having previously been discharged following treatment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients cured of cancer and are experiencing GI symptoms due to radio or chemotherapy during the last one year.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Cost of Intervention | 6 month
  The total estimated cost calculated per patient of clinical intervention for gastrointestinal problems caused by cancer treatment 1 year prior to referral to the GI and Nutrition Team. This will include number of GP visits, number and type of prescribed medicines and dietary supplements, number and type of investigations, number of visits to A&E, number of inpatient days, and number of visits from other healthcare professionals.

CONTACTS AND LOCATIONS:
Overall Officials: Jervosie Andreyev, MBBS, Phd, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom